CLINICAL TRIAL: NCT01431612
Title: The Effects of ß1-receptor Blockade and α1-adrenergic Agonist on the Kinetics of Lactated Ringer's Solution During Surgery
Brief Title: Effects of Adrenergic Drugs on the Fluid Balance During Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sodertalje Hospital (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Robert Hahn, Investigator, Sodertalje Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Esmolol study
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Ovarian Cyst
Keywords: Pharmacokinetics, kidney;; Receptors, adrenergic;; Fluids, i.v.;; Sympathetic nervous system, esmolol;; Sympathetic nervous system, phenylephrine
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esmolol (Active Comparator): 50 µg/kg/min of the ß-1-receptor-blocker esmolol (Qilu Pharmaceutical Co, Shandong, China) wss infused intravenously over 3 hours
  Interventions: Drug: Esmolol administration
- Phenylephrine (Active Comparator): Intravenous infusion of 0.01 µg/kg/min of phenylephrine (alpha1-adrenergic agonist) over 3 hours.
  Interventions: Drug: Phenylephrine infusion
- Lactated Ringer´s solution (Placebo Comparator): 10 ml/h lactated Ringer's solution without active drug was infused intravenously over 3 hours.
  Interventions: Drug: Lactated Ringer´s solution

INTERVENTIONS:
Drug: Esmolol administration — 50 µg/kg/min of the ß1-receptor-blocker esmolol was infused intravenous over 3 hours
  Other Names: Drug by Qilu Pharmaceutical Co, Shandong, China
  Arms: Esmolol
Drug: Phenylephrine infusion — 0.01 µg/kg/min of the alpha-1-adrenergic receptor agonist phenylephrine
  Other Names: Drug by Hefeng Pharmaceutical Co, Shanghai, China.
  Arms: Phenylephrine
Drug: Lactated Ringer´s solution — Intravenous Infusion of 10 ml/h lactated Ringer's solution that contained no drug
  Arms: Lactated Ringer´s solution

SUMMARY:
The aim this study was to examine to what degree the slow turnover of lactated Ringer's solution during anesthesia and surgery can be prevented by infusing esmolol (a ß1-receptor blocker) or phenylephrine in patients undergoing laparoscopic gynecological surgery performed under intravenous anesthesia.

DETAILED DESCRIPTION:
INTRODUCTION The renal clearance of infused crystalloid fluid is very low during anaesthesia and surgery, but experiments in conscious sheep indicate that the renal fluid clearance might approach a normal rate when the adrenergic balance is modified.

METHODS Sixty females (mean age, 32 years) undergoing laparoscopic gynecological surgery were randomized to control group and received only the conventional anesthetic drugs and 20 ml/kg of lactated Ringer's over 30 min. The others were also given an infusion of 50 µg/kg/min of esmolol (beta1-receptor blocker) or 0.01 µg/kg/min of phenylephrine (alpha1-adrenergic agonist) over 3 hours. The distribution and elimination of infused fluid was studied by volume kinetic analysis based on urinary excretion and blood Hgb level.

ELIGIBILITY:
Inclusion Criteria:

* ASA group I
* Scheduled for laparoscopic removal of ovarian cyst or laparoscopic hysterectomy

Exclusion Criteria:

* ASA group > I
* Daily medication

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Urinary excretion | 3 hours
  Urine was collected via an indwelling catheter during 3 hours of surgery

SECONDARY OUTCOMES:
Volume kinetics of lactated Ringer´s solution | 3 hours
  Volume kinetics was analyzed based on serial analysis of the blood Hgb concentration and the collection of urine. Distribution between a central body and a peripheral body fluid space was then calculated over time.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Hahn, MD, PhD, Principal Investigator — Södertälje Hospital, Södertälje, Sweden; Section for Anesthesia, Linköping University, Linköping, Sweden
Locations (1):
- Department of Anesthesiology, First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, China

REFERENCES:
- [Background] Vane LA, Prough DS, Kinsky MA, Williams CA, Grady JJ, Kramer GC. Effects of different catecholamines on the dynamics of volume expansion of crystalloid infusion. Anesthesiology. 2004 Nov;101(5):1136-44. doi: 10.1097/00000542-200411000-00013. PMID 15505449
- [Background] Olsson J, Svensen CH, Hahn RG. The volume kinetics of acetated Ringer's solution during laparoscopic cholecystectomy. Anesth Analg. 2004 Dec;99(6):1854-1860. doi: 10.1213/01.ANE.0000134809.07605.3C. PMID 15562086
- [Background] Ewaldsson CA, Vane LA, Kramer GC, Hahn RG. Adrenergic drugs alter both the fluid kinetics and the hemodynamic responses to volume expansion in sheep. J Surg Res. 2006 Mar;131(1):7-14. doi: 10.1016/j.jss.2005.09.012. Epub 2005 Dec 2. PMID 16325856
- [Background] Hahn RG. Volume kinetics for infusion fluids. Anesthesiology. 2010 Aug;113(2):470-81. doi: 10.1097/ALN.0b013e3181dcd88f. PMID 20613481